CLINICAL TRIAL: NCT00735163
Title: Mono-Centric, Open, Non-Controlled Study To Investigate The Feasibility Of Blood Glucose Control With The Software-Algorithm eMPC (Enhanced Model Predictive Control) In ICU Patients
Brief Title: Blood Glucose Control With A Software-Algorithm In Intensive Care Unit (ICU) Patients
Acronym: Aldea _01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Dr. Norman Kachel, B. Braun Melsungen AG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC-G-H-0806
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2009-04-16 (Estimated); Status verified 2009-04

CONDITIONS: Critical Illness
Keywords: algorithm; tight glycemic control; glucose control; intensive care; insulin; ICU
MeSH Terms: conditions — Critical Illness; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): improved model predictive control algorithm (eMPC) for glycaemic control in ICU patients
  Interventions: Other: enhanced model predictive control algorithm (eMPC)

INTERVENTIONS:
Other: enhanced model predictive control algorithm (eMPC) — eMPC (software on a bedside computer) advised insulin titration to establish tight glycaemic control

SUMMARY:
Hyperglycemia is common in critically ill patients and associated with an adverse outcome. Recently, large randomized controlled trials have demonstrated that tight glycaemic control (TGC) reduces morbidity and mortality in this population. Based on this emerging evidence intensive insulin therapy is currently finding its way into the critical care practice.

In the meantime numerous insulin infusion protocols, which are based on frequent bedside glucose monitoring, have been implemented. Recent reviews comparing different types of protocols describe widely ranging practice and difficulties in achieving TGC despite extensive efforts of the intensive care unit (ICU) staff. A fully automated algorithm may help to overcome some of these limitations by excluding intuitive interventions and integrating relevant clinical data in the decision-making process. The primary objective of the current study is to investigate the performance (efficacy) of a control algorithm for glycaemic control in ICU patients for the whole length of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years of age
* Stay in the ICU expected to be > 120 h
* Blood glucose > 110 mg/dl or patient on insulin treatment

Exclusion Criteria:

* Patients with hyperglycaemic crisis/ketoacidosis due to insulin deficiency.
* Known or suspected allergy to insulin
* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the patient (i.e., liver failure, other fatal organ failures)
* Moribund patients likely to die within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
percentage of time within the predefined glucose target range of 80-110 mg/dL | from start of treatment to the last glucose measurement under treatment

SECONDARY OUTCOMES:
hypoglycemias (lab) and possible attendant clinical symptoms (e.g. convulsions) | from start of treatment to the last glucose measurement under treatment
Usability parameters like convenience of alarming function; workload; blood sampling frequency | from start of treatment to the last glucose measurement under treatment
Concomitant medication including insulin infusion rate, parenteral/enteral nutrition | from start of treatment to the last glucose measurement under treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Pieber, Prof. Dr., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Austria

REFERENCES:
- [Background] Plank J, Blaha J, Cordingley J, Wilinska ME, Chassin LJ, Morgan C, Squire S, Haluzik M, Kremen J, Svacina S, Toller W, Plasnik A, Ellmerer M, Hovorka R, Pieber TR. Multicentric, randomized, controlled trial to evaluate blood glucose control by the model predictive control algorithm versus routine glucose management protocols in intensive care unit patients. Diabetes Care. 2006 Feb;29(2):271-6. doi: 10.2337/diacare.29.02.06.dc05-1689. PMID 16443872
- [Background] Pachler C, Plank J, Weinhandl H, Chassin LJ, Wilinska ME, Kulnik R, Kaufmann P, Smolle KH, Pilger E, Pieber TR, Ellmerer M, Hovorka R. Tight glycaemic control by an automated algorithm with time-variant sampling in medical ICU patients. Intensive Care Med. 2008 Jul;34(7):1224-30. doi: 10.1007/s00134-008-1033-8. Epub 2008 Feb 23. PMID 18297268